CLINICAL TRIAL: NCT06227624
Title: Concomitant Oral Zinc Sulfate and Phototherapy Versus Phototherapy Alone in Treatment of Neonatal Indirect Hyperbilirubinemia
Brief Title: Role of Oral Zinc in Reducing Neonatal Indirect Hyperbilirubinemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Liver Institute, Egypt (Other)
Responsible Party: Principal Investigator, Samira Abdel Wahab, Assistant professor, National Liver Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00136/2018
Record Dates: First submitted 2024-01-10; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Neonatal Jaundice
MeSH Terms: conditions — Jaundice, Neonatal | interventions — Zinc Sulfate

STUDY DESIGN:
Intervention Model Description: This randomized clinical trial was carried out on 192 neonates with indirect hyperbilirubinemia, at neonatal intensive care unit (NICU) of Pediatric Department, National Liver Institute (NLI), Menoufia University from (June 2018- June 2019). Research Ethics Committee of NLI approved the study, NLI- Institutional Review Board (IRB) protocol number is (00136/2018). Neonates enrolled in the study were randomly assigned into two groups. Group (1) (zinc and phototherapy group) included 95 neonates receiving phototherapy and oral zinc sulfate with a dose of 5 mg every 12 hours using a calibrated dropper provided with the bottle, during the period of NICU admission on phototherapy. Group (2) (phototherapy group) included 97 neonates receiving phototherapy alone. Both groups receiving phototherapy based on the guidelines of American Academy of Pediatrics for the treatment of neonatal indirect hyperbilirubinemia. Any adverse effect were noted and recorded.
Masking Description: Investigators (research staff) and parents of the patients were aware of the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- combined oral zinc salts with phototherapy (Other): neonates received combination therapy which is phototherapy and oral zinc sulfate in a dose of 5 mg every 12 hours using a calibrated dropper provided with the bottle, during the period of NICU admission of neonates on phototherapy
  Interventions: Drug: Oral zinc sulfate and standard phototherapy
- phototherapy group (No Intervention): neonates receiving phototherapy alone

INTERVENTIONS:
Drug: Oral zinc sulfate and standard phototherapy — study the role of oral zinc sulfate in reducing level of indirect hyperbilirubinemia in neonates if used with standard phototherapy
  Other Names: standard phototherapy alone
  Arms: combined oral zinc salts with phototherapy

SUMMARY:
This study aimed to determine the role of oral zinc in reducing the neonatal indirect hyperbilirubinemia if used concomitant with the standard phototherapy

DETAILED DESCRIPTION:
Unconjugated hyperbilirubinemia is one of the most common conditions in neonates. Although conventional treatment, phototherapy and/or exchange transfusion, is effective, both modalities are associated with several side effects. High levels of unconjugated hyperbilirubinemia causing direct serious brain injury, in the form of acute bilirubin encephalopathy which may progress to kernicterus (chronic bilirubin encephalopathy) with classically characterized permanently extrapyramidal movement disorders of dystonia, choreoathetosis or both, hearing loss due to auditory neuropathy spectrum, and oculomotor pareses. Treatment of unconjugated hyperbilirubinemia, such as phototherapy and blood exchange transfusion, is costly, takes a long time and can be dangerous. Phototherapy usage may associate with watery diarrhea, low serum calcium, retinal damage, skin rash, dehydration, and DNA mutation. Exchange transfusion can cause electrolyte imbalance, cardiac overload, air embolism, thrombophlebitis, thrombocytopenia, sepsis, necrotizing enterocolitis, transmission of blood-borne diseases, and portal vein thrombosis. These harmful adverse effects indicate the need to develop alternative therapeutic pharmacological strategies which aim to decrease the plasma concentration of unconjugated bilirubin by inhibiting production, stimulating hepatic clearance, or interrupting the enterohepatic circulation (EHC) of bilirubin. Studies have indicated that feeding inadequacy promotes EHC which is an important predictor for neonatal hyperbilirubinemia. Therefore, interruption of EHC is a potentially effective intervention. Various substances have been used to bind the bilirubin in intestinal lumen to prevent its absorption and disrupt enterohepatic circulation. These substances are such as oral agar, orlistat, active charcoal, cholestyramine, calcium phosphate or glucoronidase inhibitor like hydrolyzed casein; although the obtained results have been inconsistent.

Zinc is one of the critical trace elements which have a vital role in a wide range of biological activities in living organisms. Mendez-Sanchez et al., 2001 study was the first one which reported that zinc salts at physiological fluid media can be flocculated and almost completely adsorb unconjugated bilirubin from unsaturated micellar bile salt solutions. Vitek et al., 2005 studied the effect of zinc salts ingestion in hyperbilirubinemic rats and reported that oral zinc salts can decrease serum bilirubin levels efficiently, due to the probable enterohepatic circulation inhibition of bilirubin. Méndez-Sánchez et al., 2022 showed that administration of oral zinc sulphate can significantly decrease serum indirect bilirubin levels in adult patients with Gilbert´s syndrome.

Therefore, the anticipated role of zinc supplementation in neonatal jaundice seems to be an attractive issue for research. This study aimed to determine the role of oral zinc on treatment of neonates suffering from unconjugated hyperbilirubinemia with variable gestational ages, different levels of jaundice severity and different birth weight.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with total serum bilirubin (TSB) exceeding the 40th percentile track for age as per the hour-specific bilirubin nomogram of the American Academy of Pediatrics (AAP)
* Neonates who have indirect hyperbilirubinemia, not indicated for exchange transfusion.

Exclusion Criteria:

* Neonates submitted to blood transfusion.
* Neonates indicated for exchange transfusion
* Associated congenital anomalies.
* Co-morbidities such as sepsis, pneumonia or respiratory distress.
* Neonates whom their mothers received phenobarbitone during the third trimester

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Determine the role of oral zinc in reducing level of unconjugated hyperbilirubinemia | Baseline
  Measurement of serum bilirubin after receiving zinc/ phototherapy and phototherapy alone

CONTACTS AND LOCATIONS:
Overall Officials: Heba S. Sallam, specialist, Principal Investigator — Al-Dalangat Central Hospital, Beheira, Egypt; Hala H. Elsaeed, professor, Study Chair — National liver institute. Menoufia university, Egypt; Mohsen H Hussein, professor, Study Chair — National liver institute. Menoufia university, Egypt; Hanaa A. El- Alraby, Study Director — National liver institute. Menoufia university, Egypt
Locations (1):
- National Liver Institute, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
tabulated data in results of full perinatal and maternal history including maternal age, parity, and presence of jaundice in previous sibling were collected for all neonates. Routine general and systemic examination, laboratory investigations including complete blood count, reticulocytic count, C-reactive protein, ABO blood grouping and Rh type for neonates and their mothers and neonatal serum zinc level on admission to NICU were done. Measurement of TSB and DSB were done on admission and serially according to case severity and response to treatment, until discharge then after 24 and 72 hours after stoppage of phototherapy to detect rebound hyperbilirubinemia.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after research submission, and for ever
Access Criteria: journal web sit of publication

REFERENCES:
- [Background] • Kumar A, Bagri NK, Basu S, Asthana RK. Zinc Supplementation for Neonatal Hyperbilirubinemia: A Randomized Controlled Trial. Indian Pediatrics . 2014; 51:375-378. • Watchko JF, Tiribelli C. Bilirubin-Induced Neurologic Damage- Mechanisms and Management Approaches. New England Journal of Medicine. 2013; 369:2021-2030. • Olusanya B O, Imam Z O, Emokpae A A, Iskander IF. Revisiting the criteria for exchange transfusion for severe neonatal hyperbilirubinemia in resource-limited settings. Neonatology. 2016; 109:97-104. • Cuperus F, Hafkamp A, Hulzebos C, Verkade H. Pharmacological therapies for unconjugated hyperbilirubinemia. Current pharmaceutical design. 2009; 15:2927-2938. • Prashanth GP. The Significance of Enterohepatic Circulation in the Causation Neonatal Hyperbilirubinemia. The Indian Journal of Pediatrics. 2012; 79:1251-1252. • Patil R, Sontakke T, Biradar A, Nalage D. Zinc: an essential trace element for human health and beyond. Food and Health. 2023; 5(3):13.
- [Background] • Méndez-Sánchez N, Roldán-Valadez E, Flores M A, Cárdenas-Vázquez R, Uribe M. Zinc salts precipitate unconjugated bilirubin in vitro and inhibit enterohepatic cycling of bilirubin in hamsters. Eur J Clin Invest. 2001; 31(9):773-80. • Vitek L, Muchova L, Zelenka J, et al. The effect of zinc salts on serum bilirubin levels in hyperbilirubinemic rats. J Pediatr Gastroenterol Nutr. 2005; 40:135-140. • Méndez-Sánchez N, Martínez M, González V, Roldán-Valadez E, Flores M A Uribe M. Zinc sulfate inhibits the enterohepatic cycling of unconjugated bilirubin in subjects with Gilbert's syndrome. Annals of hepatology. 2022; 1(1): 40-43 • Bhutani VK, Johnson L, Sivieri EM. Predictive Ability of a Predischarge Hour-specific Serum Bilirubin for Subsequent Significant Hyperbilirubinemia in Healthy Term and Near-term Newborns. Pediatrics. 1999; 103:6-14.
- [Background] • Duryea EL, Hawkins JS, McIntire DD, Casey BM, Leveno KJ. A Revised Birth Weight Reference for the United States. Obstetrics & Gynecology. 2014; 124. • Rasul CH, Hasan MA, Yasmin F. Outcome of neonatal hyperbilirubinemia in a tertiary care hospital in bangladesh. The Malaysian journal of medical sciences: MJMS. 2010; 17:40-44. • Johnsen Ø, Eliasson R. Evaluation of a commercially available kit for the colorimetric determination of zinc in human seminal plasma. International Journal of Andrology. 1987; 10:435-440. • Rana N, Mishra S, Bhatnagar S, Paul V, Deorari AK, Agarwal R. Efficacy of Zinc in Reducing Hyperbilirubinemia among At-Risk Neonates: A Randomized, Double-Blind, Placebo-Controlled Trial. The Indian Journal of Pediatrics. 2011; 78:1073-1078. • Patton P, Rachmadi D, Sukadi A. Effect of oral zinc on hyperbilirubinemia in full term neonates. Paediatrica Indonesiana. 2011; 51:107-10. • Faal G, Masjedi HK, Sharifzadeh G, Kiani Z. Efficacy of zinc sulfate on indirect hyperbilirubinemia in premature infants admitted to neonatal intensive care unit: a double-blind, randomized clinical trial. BMC pediatrics. 2020; 20:1-7.
- [Background] • Mandlecha TH, Mundada SM, Gire PK, Reddy N, Khaire P, Joshi T, Pawar S. Effect of Oral Zinc Supplementation on Serum Bilirubin Levels in Term Neonates With Hyperbilirubinemia Undergoing Phototherapy: A Double-blind Randomized Controlled Trial. Indian Pediatrics. 2023; 60:991-995. • Elfarargy MS, Al-Ashmawy MG, Abu-Risha SE, Khattab H. Zinc Supplementation in Preterm Neonates with Jaundice: Is it Beneficial?. Endocr Metab Immune Disord Drug Targets. 2021; 21(10):1929-1934. • Mafinezhad S, Bayani G, Bozorgnia Y, Khodaparast M, Jodat S. Effect of oral zinc sulfate on reducing hyperbilirubinemia among newborns under 1800 gram. Journal of North Khorasan University of Medical Sciences. 2016; 7:897-904. • Indrio F, Baldassarre ME, Francavilla R. Will Hyperbilirubinemic Neonates Ever Benefit from Oral Zinc Salt?. Journal of Pediatric Gastroenterology and Nutrition. 2006; 42:118-119.